CLINICAL TRIAL: NCT04518683
Title: Evaluation of a New Treatment Using Mobile Applications in the Treatment of Stress Urinary Incontinence in Women Outside the Peripartum - Pilot Study
Brief Title: Rehabilitation With Mobile Applications in Women With SUI
Acronym: SUI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences of Western Switzerland (Other)
Collaborators: Claire de Labrusse (Unknown); Sandrine Balisson (Unknown); Léa Dassonville (Unknown)
Responsible Party: Principal Investigator, Bertuit Jeanne, Professor Associated, University of Applied Sciences of Western Switzerland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-01978
Record Dates: First submitted 2020-08-12; First posted 2020-08-19 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Urinary Incontinence; Stress Urinary Incontinence
Keywords: stress urinary incontinence; mobile application; woman
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: study pilot mixte by a quantitative part corresponding to a randomized controlled intervention study and a phenomenological qualitative aspect
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Free randomization via a pre-established listing including a coding system (0-intervention group and 1-control group) will be set up. A set of 30 opaque envelopes including a coding will be drawn for each participant by a person other than the principal investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Groupe 1 - Study group (Experimental): The home program (outside of the sessions with the physiotherapist) will be done with a mobile application equipped with a vaginal probe. The exercises should be done 3x/week for 10 minutes (time corresponding to 1 programe). The correct use of the prob will have been checked during the sessions with the physiotherapist. This training will work on the strength, relaxation and endurance of the pelvic floor.
  The program includes 3 levels of difficulty. Once the user has successfully completed one level, she can move on to the next.
  Interventions: Device: Perineal rehabilitation with mobile applications for women with SUI
- Groupe 2 - Control group (Active Comparator): The home program (outside of the sessions with the physiotherapist) will be done without a mobile application. The exercises will have been explained during the sessions with the physiotherapist by oral instructions. The exercises will be done 3x/week for 10 minutes. The correct realization of the exercises will have been verified during the sessions with the physiotherapist.
  This training will work on pelvic floor strength, relaxation and endurance. The program includes 3 levels of difficulty
  Interventions: Device: Classic perineal rehabilitation for women with SUI

INTERVENTIONS:
Device: Perineal rehabilitation with mobile applications for women with SUI — Physiotherapy: Sessions with the physiotherapist will consist of information on anatomy, perineal awareness and behavioural therapy. The therapist will educate the patient on pelvic floor contraction/relaxation. the sessions will remain personalized and standardized like a classic treatment, and will also aim to work on motivation. 9 sessions during 3 months.
  Home Program: The home program will be done with a mobile application equipped with a vaginal probe. The exercises should be done 3x/week for 10 minutes. The correct use of the prob will have been checked during the sessions with the physiotherapist. This training will work on the strength, relaxation and endurance of the pelvic floor.The program includes 3 levels of difficulty. Once the user has successfully completed one level, she can move on to the next.
  Arms: Groupe 1 - Study group
Device: Classic perineal rehabilitation for women with SUI — Physiotherapy: Sessions with the physiotherapist will consist of information on anatomy, perineal awareness and behavioural therapy. The therapist will educate the patient on pelvic floor contraction/relaxation. The sessions will remain personalized and standardized like a classic treatment, and will also aim to work on motivation. 9 sessions during 3 months.
  Home program: The home program will be done without a mobile application. The exercises will have been explained during the sessions with the physiotherapist by oral instructions. The exercises will be done 3x/week for 10 minutes. The correct realization of the exercises will have been verified during the sessions with the physiotherapist.
  Arms: Groupe 2 - Control group

SUMMARY:
Stress urinary incontinence (SUI) is the most common form of urinary incontinence in women. It affects women in their quality of life : physical, social, sexual and psychological levels. International recommendations suggest conservative treatments as first-line by training the pelvic floor muscles with or without a biofeedback-type control system. The latter allows the patient to visualize her muscle activity while stimulating her motivation. The part of adherence and compliance is very important in this rehabilitation where the woman must provide a significant commitment to continue the exercises beyond the support of the physiotherapist. In this area, a new approach is emerging with the arrival of health applications on smartphones. However, these tools lack scientific validation. The objective of this mixed pilot study (randomized controlled study with a qualitative part) is to investigate a new treatment for middle-aged to advanced patients outside the period of peripartum suffering from SUI, through an application mobile with probe as home program in standard physiotherapist treatment.

DETAILED DESCRIPTION:
The quantitative component is composed of 2 arms and the intervention is during 3 months:

* Study group : half of the participants will have a home pelvic floor work program via a mobile application in addition to therapeutic follow-up by a physiotherapist.
* Control group: the other half will perform the home pelvic floor work program without application and will also have therapeutic follow-up by a physiotherapist.

The qualitative component will include individual and semi-structured interviews based on an interview guide with 4 women in the study group and 4 women in the other group after completion of their perineal rehabilitation program.

The protocol will be offered to patients who meet the inclusion criteria (see below). Participants will be randomized into one of the two groups using sealed opaque envelopes, the order of which will have been randomly generated by randomization software.

Recruitment of participants will be done with the help of partner doctors. They will be responsible for introducing them to the study and providing them with the necessary documentation (information and informed consent sheets, 9 physiotherapy sessions for the treatment of SUI and the list of physiotherapists from the ASPUG-PP adapted to the study). The physiotherapists included in this study are all specialized in pelvi-perineology and members of ASPUG-PP and trained in the study protocol. They will ensure running of the process by collecting information from the anamnesis and carrying out pre- and post-tests with the project team.

The data will be entered directly by the investigator or one of the collaborators in Redcap. All information required by the protocol should be entered as it is obtained and an explanation should be provided for any missing data. Data analysis will be performed with the intention of addressing the study design. A drop-out rate of 30% is taken into account in the calculation of the sample size.

The sample size was estimated based on the ICQI-SF (intensity of UI symptoms) data from the study by Asklund et al (2018) because these are the only data available for an accurate calculation. The probability of error (alpha) was set at 0.10 and the power (1-beta) at 0.95. Based on these values, the sample size was calculated at 30 participants, or 15 per group. The standard deviation considered is 3.5 and the desired effect size is d=0.8 (strong).

Descriptive statistics will be carried out on the feasibility outcomes and on the outcomes of the final trial. Intention-to-treat analysis, inferential statistics will be considered in order to obtain primary results from the final trial. The objective is to investigate the relevance of the project by assessing differences between groups (inter-group analysis) and between evaluations (intra-group analysis). The thematic analysis of the qualitative data will be carried out in four phases as described by Braun & Clarke (2006) : (1) familiarization (2) identification of themes and units of meaning; (3) coding of transcripts; (4) concordance and reduction of redundancies. Phase 4 will allow for the comparison of categories and their refinement. The thematic analysis has the advantage of highlighting the analysis process through its transparency and the links between the stages of analysis.

ELIGIBILITY:
Inclusion Criteria:

* women with SUI diagnosed by a doctor

Exclusion Criteria:

* Post-partum at least 1 year
* pregnant women
* mixt urinary incontinence

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Acceptability of study with information from doctor, physiotherapist and patients | 6 months
  Number of patients with the eligibility criteria over the recruitment period , Number of patients contacting physiotherapists to participate in the study over the recruitment period - Number of patients signing informed consent, enrolled over the duration of the study.
  Number of dropouts, timing. For each participant: her follow-up with dates. The patient's satisfaction with the PGI-I (Patient Global Impression Improvement). This questionnaire will be completed at the post-test observance of design: it will be evaluated via a "logbook" distributed to the patient . In relation to feasibility, we will evaluate the following parameters: The number of participants who complete the diary - The number of participants who follow the study guidelines - The number of participants who complete the home program, how often, for how long The number of participants who agree to participate in interviews

SECONDARY OUTCOMES:
Adherence - Incontinence Treatment Motivation Questionnaire (ITMQ) | 3 months
  via the Incontinence Treatment Motivation Questionnaire (ITMQ) pre- and post-tests performed during appointments with the partner physiotherapist. The questionnaires will be completed by the project team with the participant.
Observance- logbook | 3 months
  it will be evaluated via a "logbook" distributed to the patient to indicate the completion of the home program on a daily basis.
IU symptom - International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF)- urinary calenda | 3 months
  via the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) and a urinary calendar. The latter must be completed over 3 days at the beginning (pre-test) and end (post-test) of each participant's care.
Pelvic floor muscle functionality - PERFECT | 3 months
  via PERFECT (P-power or pressure, E-endurance, R-repetition, F-fast contractions, ECT- every contraction timed) using digital vaginal palpation and the modified Oxford scale. pre- and post-tests performed during appointments with the partner physiotherapist. The questionnaires will be completed by the project team with the participant.
Quality of life - DITROVIE | 3 months
  via DITROVIE. pre- and post-tests performed during appointments with the partner physiotherapist. The questionnaires will be completed by the project team with the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Bertuit, PhD, Principal Investigator — University of Applied Sciences of Western Switzerland
Locations (1):
- Bertuit, Lausanne, Canton of Vaud, Switzerland